CLINICAL TRIAL: NCT06128356
Title: Pilot Study of Dexmedetomidine Sublingual Film for the Ambulatory Treatment of Hyperadrenergic Autonomic Crisis in Patients With Familial Dysautonomia
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-00174
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Familial Dysautonomia
MeSH Terms: conditions — Dysautonomia, Familial | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sublingual dexmedetomidine (Experimental): Participants will be administered two 60 micrograms sublingual films of IGLMI following start of an autonomic crises. The maximum amount for the study is four oral films of 60 micrograms in 24 hours, two at the beginning of the crises and if needed, two additional within two hours.
  Interventions: Drug: Dexmedetomidine Sublingual

INTERVENTIONS:
Drug: Dexmedetomidine Sublingual — Dexmedetomidine 120 mcg on two thin dissolvable films for sublingual administration
  Other Names: IGALMI

SUMMARY:
This is a pilot open-label study to evaluate the feasibility of conducting a clinical trial using sublingual dexmedetomidine sublingual film to treat hyperadrenergic autonomic crises in patients with Familial Dysautonomia at home. The primary aims are to examine the feasibility of performing a clinical trial using dexmedetomidine at home to terminate autonomic crisis, and refine the interventions and assessments used to evaluate autonomic crisis termination.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed diagnosis of Familial Dysautonomia.
* Evidence of autonomic crisis, previous treatment with IV dexmedetomidine without significant side effects, and registered medical data within the year preceding the study in our database.
* One or more autonomic crises during the last year.
* Age above 18 years.
* The patient has a responsible caretaker to communicate with the medical providers.
* Provision of signed and dated informed consent form from the patient and responsible caregiver.
* Able to state willingness to comply with all study procedures and availability for the duration of the study
* For males and females of reproductive potential: use condoms for contraception if sexually active.

Exclusion Criteria:

* At the consideration of the principal investigator, the caregiver cannot fully understand the protocol or communicate during the crisis with the Center.
* The patient during the crisis, before taking the medication, has any of the following:
* a. Oxygen saturation less than 92% on room air or baseline need for oxygen, change from baseline oxygen dependency.
* b. Respiratory rate >20 breaths per minute.
* c. Supine blood pressure ≤ 90/60mmHg
* d. Febrile illness with temperature >100.3 F.
* e. Serological signs of infection (WBC count >10 g/dL, or CRP >10 mg/L or ESR>20, or above their steady historical baseline levels) in recent (less than one month) studies.
* The patient is a female and has a positive pregnancy test.
* MoCA score <25 points.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects screened per month | Month 6
Number of subjects enrolled per month | Month 6
Number of completed crises treated at home within the protocol | Month 6
Number of subjects that underwent an autonomic crisis per month | Month 6
Average duration of the study from visit 1 to the last visit of the last patient | From enrollment to end of treatment (up to 6 months)

SECONDARY OUTCOMES:
Length of time from autonomic crisis onset to the initiation of the video recording | Up to 2 hours
Length of time from autonomic crisis onset to administration of the medication | Up to 2 hours
Length of time from autonomic crisis onset to crisis resolution | Up to 24 hours
Length of time it took to complete assessments from start of autonomic crisis | Up to 24 hours
Percentage of completion of all rating scales | Month 6
  The scales required to be completed is the Autonomic Crisis Symptom Assessment Scale (ACSAS), the study safety assessments and the Richmond Agitation-Sedation Scale.
Change in blood pressure | Pre-dose, up to 2 hours post-dose
Change in heart rate | Pre-dose, up to 2 hours post-dose
Change in number of vomiting episodes | Pre-dose, up to 2 hours post-dose
Change in number of retching episodes | Pre-dose, up to 2 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Gonzalez-Duarte, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Alejandra.gonzalez-duarte@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be provided access upon reasonable request. Requests should be directed to Alejandra.gonzalez-duarte@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.